CLINICAL TRIAL: NCT03298373
Title: 28-Day Repeat-Dose, Dose Escalation Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics Study of 11-β Methyl Nortestosterone Dodecylcarbonate (11β-MNTDC) in Healthy Men
Brief Title: 28-Day Repeat-Dose, Dose Escalation Study of 11-β Methyl Nortestosterone Dodecylcarbonate (11β-MNTDC) in Healthy Men
Acronym: CCN014A
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CCN014A
Record Dates: First submitted 2017-09-22; First posted 2017-10-02 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Healthy Men; Male Contraception
Keywords: Healthy Men; Male Contraception; Androgen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsules that look like the 11β-MNTDC capsules but with no active ingredients.
  Interventions: Drug: Placebo
- 11β-MNTDC (Experimental): 11β-MNTDC capsules administered orally (200 mg or 400 mg).
  Interventions: Drug: 11β-methyl-nortestosterone-dodecylcarbonate

INTERVENTIONS:
Drug: Placebo — Placebo capsules that look like the 11β-MNTDC capsules but with no active ingredients.
  Arms: Placebo
Drug: 11β-methyl-nortestosterone-dodecylcarbonate — 11β-MNTDC doses in castor oil/benzyl benzoate capsules (100 mg each) administered in 200 mg or 400 mg doses orally.
  Arms: 11β-MNTDC

SUMMARY:
This is a Phase I multicenter, double-blind, repeat dose, dose-escalating study, in healthy men to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics of 11-β Methyl Nortestosterone Dodecylcarbonate (11β-MNTDC).

DETAILED DESCRIPTION:
This repeat dose, dose-ranging study will be conducted at two centers: the Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center and the University of Washington.

Two doses of 11β-MNTDC (200 mg and 400 mg) were selected for a dose-escalating 28-day repeat dose study. Twenty subjects will complete this study at each of the 11β-MNTDC (15 on 11β-MNTDC and 5 on placebo) yielding a total of 40 completed subjects (30 on 11β-MNTDC and 10 on placebo) across both sites. Safety will be assessed in subjects receiving the lower dosage before additional men receive the higher dose for 28 days. In addition to safety and tolerability, suppression of serum T, calculated free T, E2, gonadotropins (LH & FSH), and SHBG will also be assessed as secondary pharmacodynamic (PD) endpoints. The 24-hour detailed PK of 11β-MNTDC will be assessed on Days 1 and 28. Trough levels of 11β-MNTDC will be obtained throughout the 28-day treatment period, at 48 and 72 hours (Days 30 and 31) after the last dose and at the End of Study visit (between Days 70-76).

ELIGIBILITY:
Inclusion Criteria:

Men who meet all the following criteria are eligible for enrollment in the trial:

1. Male volunteers in good health as confirmed by physical examination, medical history, and clinical laboratory tests of blood and urine at the time of screening.
2. 18 to 50 years of age (inclusive) at the time of the enrollment visit.
3. BMI ≤ 33 calculated as weight in kg/ (height in m2).
4. No history of hormonal therapy use in the three months prior to the first screening visit.
5. Subject agrees to use a recognized effective method of contraception with any female partner during the course of the study.
6. Subjects agrees to refrain from donating blood or plasma during the study period and from participating in other investigational drug studies.
7. Subjects agrees to refrain from excessive alcohol consumption during the study period. (No more than 15 drinks per week and no alcohol consumption within 24 hours of a study visit.)
8. Subjects agrees to refrain from significant changes in their current exercise regimen during the drug exposure period.
9. No known or suspected current alcohol dependence syndrome, chronic marijuana use, or any illicit drug use that may affect metabolism/transformation of steroid hormones and study treatment compliance.
10. In the opinion of the investigator, subject can comply with the protocol, understand and sign an informed consent and HIPAA form.

Exclusion Criteria:

Men who meet any of the following criteria are NOT eligible for enrollment in the trial:

1. Men participating in another clinical trial involving an investigational drug within 30 days prior to the first screening visit.
2. Men not living in the catchment area of the clinic or within a reasonable distance from the study site.
3. Clinically significant abnormal physical or laboratory findings at screening.
4. Elevated PSA (levels ≥ 2.5 ng/mL) at screening, per local laboratory normal values.
5. Abnormal serum chemistry values at screening, per local laboratory reference ranges that indicate liver or kidney dysfunction or that may be considered clinically significant. In addition, the following upper limits will be observed: fasting bilirubin less than 2 mg/dL, cholesterol less than 221 mg/dL, and fasting triglycerides less than 201 mg/dL.
6. Abnormal semen analyses or abnormal semen concentration as defined by the WHO semen manual.
7. Use of androgens within 3 months before the first screening visit except for long acting, intramuscular testosterone undecanoate which will require a wash out period of 6 months prior to randomization.
8. Ongoing use of body building substances including nutritional supplements.
9. Systolic BP > 135 mm Hg and Diastolic blood pressure BP > 85 and mm Hg; Blood pressure (BP) will be taken 3 times at 5 - minute intervals and the mean of all measurements be used to determine eligibility.
10. Clinically significant abnormal EKG or a QTc interval of > 450 msec.
11. PHQ-9 score of 15 or above.
12. History of hypertension, including hypertension controlled with medication.
13. Known history of primary testicular disease or disorders of the hypothalamic-pituitary axis.
14. Benign or malignant liver tumors, active liver disease or known non-alchoholic fatty liver disease (NAFLD)
15. History of breast carcinoma.
16. Known history of androgen deficiency due to hypothalamic-pituitary or testicular disease.
17. Known history of cardiovascular, renal, hepatic or prostatic disease or significant psychiatric illness.
18. Positive serology for active Hepatitis (not immunization-related serology) or HIV at screening visit.
19. A serious systemic disease such as diabetes mellitus.
20. History of known, untreated sleep apnea.
21. Partner is known to be pregnant.
22. Men desiring fertility within the first 24 weeks of study participation.
23. Men participating in competitive sports where drug screening for prohibited substances (including anabolic steroids) is routine. Exclusion is due to the potential of testing positive for androgens that may occur from their study participation coupled with the unknown efficacy (i.e. duration of positive testing) of a single dose.
24. Subjects taking anticonvulsants.
25. Subjects taking recombinant human growth factor (HGH).
26. Subjects with a hematocrit greater than 55%.
27. Previous participation in this clinical trial or any trials of 11-Beta MNTDC.
28. Any site staff member with delegated study responsibilities or a family member of a site staff member with delegated study responsibilities.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 43 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2020-02-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (safety and tolerability) of repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in sodium (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in postassium (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in chloride (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in bicarbonate (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in fasting glucose (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in creatinine (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in calcium (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in total bilirubin (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in alkaline phosphatase (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in alanine aminotransferase (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in aspartate transaminase (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in albumin (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in blood urea nitrogen (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in body mass index (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in blood pressure (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in pulse (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in respiratory rate (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days
Changes from baseline in QTc interval (safety and tolerability) with repeated daily oral dosing of 11β-MNTDC. | 28 days

SECONDARY OUTCOMES:
Pharmacokinetics of 11β-MNTDC using AUC (0-24). | 28 days
Pharmacodynamics of 11β-MNTDC by assessing the suppression of serum Testosterone (T) using mean values at each visit. | 28 days
Pharmacodynamics of 11β-MNTDC by assessing the suppression of Estradiol (E2) using mean values at each visit. | 28 days
Pharmacodynamics of 11β-MNTDC by assessing the suppression of Follicle Stimulating Hormone (FSH) using mean values at each visit. | 28 days
Pharmacodynamics of 11β-MNTDC by assessing the suppression of Luteinizing Hormone (LH) using mean values at each visit | 28 days
Pharmacodynamics of 11β-MNTDC by assessing the suppression of Sex Hormone Binding Globulin (SHBG) using mean values at each visit. | 28 days
Changes from baseline in sexual function (safety and tolerability) with 11β-MNTDC after 28 days of dosing using the psychosexual daily questionnaire. | 28 days
Changes from baseline in mood (safety and tolerability) with 11β-MNTDC after 28 days of dosing using the Patient Health Questionnaire-9. | 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Washington Medical Center & Health Sciences, Seattle, Washington